CLINICAL TRIAL: NCT00389597
Title: LDR Spine USA Mobi-C(R) Cervical Disc Prosthesis IDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LDR Spine USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LDR-001
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Degenerative Disc Disease
Keywords: degenerative disc disease; cervical arthroplasty; Mobi C; multilevel; anterior cervical discectomy and fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Level (Experimental): Cervical artificial disc (investigational device) at 1 level compared with control procedure (ACDF) at one level
  Interventions: Device: Cervical Artificial Disc
- 2 Level (Experimental): Cervical artificial disc (investigational device) at 2 levels compared with control procedure (ACDF) at two levels
  Interventions: Device: Cervical Artificial Disc

INTERVENTIONS:
Device: Cervical Artificial Disc — Cervical artificial disc mechanical device

SUMMARY:
The purpose of this investigation is to establish the safety and effectiveness of the LDR Spine Mobi-C® Cervical Disc Prosthesis which is an anterior cervical interbody mechanical device. The primary objective of the study is to evaluate the overall success rate of the investigational device as compared to the control in the treatment of patients with symptomatic DDD with radiculopathy or myeloradiculopathy at one or two adjacent levels. Patients should be without prior cervical fusion between C3 and C7 and unresponsive to non-operative conservative treatment for six weeks after symptom onset or have the presence of progressive symptoms or signs of nerve/spinal cord compression despite continued non-operative conservative treatment.

DETAILED DESCRIPTION:
Objectives of the Investigation

The purpose of this investigation is to establish the safety and effectiveness of the LDR Spine Mobi-C® Cervical Disc Prosthesis which is an anterior cervical interbody mechanical device. The primary objective of the study is to evaluate the overall success rate of the investigational device as compared to the control in the treatment of patients with symptomatic DDD with radiculopathy or myeloradiculopathy at one or two adjacent levels. Patients should be without prior cervical fusion between C3 and C7 and unresponsive to non-operative conservative treatment for six weeks after symptom onset or have the presence of progressive symptoms or signs of nerve/spinal cord compression despite continued non-operative conservative treatment.

Study Design Rationale

The study is a prospective, randomized, multi-center, concurrently controlled investigation, in which the study device will be compared to the control treatment consisting of conventional anterior cervical discectomy and fusion (ACDF) in accordance with the Smith-Robinson procedure. Patients will be followed for two years postsurgery (primary endpoint) and at 3, 4, 5, and 7 years thereafter.

Duration of the Investigation

Patients will be followed post-operatively at 6 weeks, and 3-, 6-, 12-, 18-, and 24-months. After 24 months, patients will continue to be followed at 3,4, 5 and 7 years.

Design Techniques to Avoid Bias

To eliminate selection bias, investigational and control comparison groups will be assigned at random.

Institutional Review Board

No clinical studies will begin without documented approval of the clinical investigation by the Institutional Review Board (IRB) affiliated with the study center.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-69 years.
2. Diagnosis of radiculopathy or myeloradiculopathy of the cervical spine, with pain, paresthesias or paralysis in a specific nerve root distribution C3 through C7, including at least one of the following:

   * Neck and/or arm pain (at least 30mm on the 100mm VAS scale).
   * Decreased muscle strength of at least one level on the clinical evaluation 0 to 5 scale.
   * Abnormal sensation including hyperesthesia or hypoesthesia; and/or
   * Abnormal reflexes
3. Symptomatic at one or two adjacent levels from C3 to C7;
4. Radiographically determined pathology at one or two adjacent level(s) to be treated correlating to primary symptoms including at least one of the following:

   * Decreased disc height on radiography, CT, or MRI in comparison to a normal adjacent disc.
   * Degenerative spondylosis on CT or MRI.
   * Disc herniation on CT or MRI;
5. Neck Disability Index Score of ≥15/50 or ≥30%;
6. Unresponsive to non-operative, conservative treatment (rest, heat, electrotherapy, physical therapy, chiropractic care and/or analgesics) for:

   * Approximately six weeks from radiculopathy or myeloradiculopathy symptom onset; or
   * Have the presence of progressive symptoms or signs of nerve root/spinal cord compression despite continued non-operative conservative treatment.

Note: Not a complete listing

Exclusion Criteria:

1. Reported to have an active systemic infection or infection at the operative site;
2. Reported to have a history of or anticipated treatment for active systemic infection, including HIV or Hepatitis C;
3. More than one immobile vertebral level between C1 to C7 from any cause including but not limited to congenital abnormalities and osteoarthritic "spontaneous" fusions;
4. Previous trauma to the C3 to C7 levels resulting in significant bony or disco-ligamentous cervical spine injury;
5. Reported to have had any prior spine surgery at the operative level;
6. Reported to have had prior cervical fusion procedure at any level;
7. Axial neck pain in the absence of other symptoms of radiculopathy or myeloradiculopathy justifying the need for surgical intervention;
8. Disc height less than 3mm as measured from the center of the disc in a neutral position and disc height less than 20% of the anterior-posterior width of the inferior vertebral body;
9. Radiographic confirmation of severe facet joint disease or degeneration;

Note: Not a complete listing

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2006-04; Primary Completion 2010-03 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Rashbaum, MD, Principal Investigator — Texas Back Institute
Locations (24):
- United States (24):
  - Texas Back Institute-West, Phoenix, Arizona
  - Southern California Institute of Neurological Surgery, Escondido, California
  - Massoudi & Jackson Neurosurgical Association, Laguna Hills, California
  - Memorial Orthopaedic Surgical Group, Long Beach, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - University of California- Davis Medical Center, Sacramento, California
  - Spine Institute at St. John's Health Center, Santa Monica, California
  - Stanford University, Stanford, California
  - Panorama Orthopedics and Spine Care, Golden, Colorado
  - Southeastern Clinical Research, Orlando, Florida
  - Orthopaedics North East, Fort Wayne, Indiana
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - GBMC Healthcare, Baltimore, Maryland
  - University Neurologic Systems, Detroit, Michigan
  - St. Mary's of Saginaw Field Neurosciences Institute, Saginaw, Michigan
  - Simmons Orthopaedics and Spine Associates, Buffalo, New York
  - Orthopedic Spine Care of Long Island, Melville, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - Oklahoma Spine & Brain Institute, Tulsa, Oklahoma
  - Austin Brain and Spine, Austin, Texas
  - Foundation Surgical Hospital, Houston, Texas
  - West Texas Spine, Odessa, Texas
  - Texas Back Institute, Plano, Texas
  - Texas Spine and Joint Hospital, Tyler, Texas

REFERENCES:
- [Result] Hisey MS, Bae HW, Davis R, Gaede S, Hoffman G, Kim K, Nunley PD, Peterson D, Rashbaum R, Stokes J. Multi-center, prospective, randomized, controlled investigational device exemption clinical trial comparing Mobi-C Cervical Artificial Disc to anterior discectomy and fusion in the treatment of symptomatic degenerative disc disease in the cervical spine. Int J Spine Surg. 2014 Dec 1;8:7. doi: 10.14444/1007. eCollection 2014. PMID 25694918
- [Result] Davis RJ, Kim KD, Hisey MS, Hoffman GA, Bae HW, Gaede SE, Rashbaum RF, Nunley PD, Peterson DL, Stokes JK. Cervical total disc replacement with the Mobi-C cervical artificial disc compared with anterior discectomy and fusion for treatment of 2-level symptomatic degenerative disc disease: a prospective, randomized, controlled multicenter clinical trial: clinical article. J Neurosurg Spine. 2013 Nov;19(5):532-45. doi: 10.3171/2013.6.SPINE12527. Epub 2013 Sep 6. PMID 24010901
- [Derived] Radcliff K, Davis RJ, Hisey MS, Nunley PD, Hoffman GA, Jackson RJ, Bae HW, Albert T, Coric D. Long-term Evaluation of Cervical Disc Arthroplasty with the Mobi-C(c) Cervical Disc: A Randomized, Prospective, Multicenter Clinical Trial with Seven-Year Follow-up. Int J Spine Surg. 2017 Nov 28;11(4):31. doi: 10.14444/4031. eCollection 2017. PMID 29372135
- [Derived] Radcliff K, Coric D, Albert T. Five-year clinical results of cervical total disc replacement compared with anterior discectomy and fusion for treatment of 2-level symptomatic degenerative disc disease: a prospective, randomized, controlled, multicenter investigational device exemption clinical trial. J Neurosurg Spine. 2016 Aug;25(2):213-24. doi: 10.3171/2015.12.SPINE15824. Epub 2016 Mar 25. PMID 27015130
- [Derived] Jackson RJ, Davis RJ, Hoffman GA, Bae HW, Hisey MS, Kim KD, Gaede SE, Nunley PD. Subsequent surgery rates after cervical total disc replacement using a Mobi-C Cervical Disc Prosthesis versus anterior cervical discectomy and fusion: a prospective randomized clinical trial with 5-year follow-up. J Neurosurg Spine. 2016 May;24(5):734-45. doi: 10.3171/2015.8.SPINE15219. Epub 2016 Jan 22. PMID 26799118
- [Derived] Davis RJ, Nunley PD, Kim KD, Hisey MS, Jackson RJ, Bae HW, Hoffman GA, Gaede SE, Danielson GO 3rd, Gordon C, Stone MB. Two-level total disc replacement with Mobi-C cervical artificial disc versus anterior discectomy and fusion: a prospective, randomized, controlled multicenter clinical trial with 4-year follow-up results. J Neurosurg Spine. 2015 Jan;22(1):15-25. doi: 10.3171/2014.7.SPINE13953. PMID 25380538
- See also: FDA Approval 2 Level — https://www.accessdata.fda.gov/cdrh_docs/pdf11/P110009A.pdf
- See also: FDA Approval 1 Level — https://www.accessdata.fda.gov/cdrh_docs/pdf11/P110002A.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One Level TDR Arm: 169 subjects randomized (5 not operated) One Level ACDF Arm: 87 subjects randomized (6 not operated) Two level TDR arm: 232 subjects randomized (7 not operated). Two Level ACDF Arm: 115 subjects randomized (10 not operated)
Pre-assignment Details: 1 level TDR enrolled 184 incl15 training cases (2 withdrew consent, 1 AE, 2 other). 1 level ACDF enrolled 87 with no training cases (4 withdrew consent, 2 other) for 245 randomized subjects. 2 level TDR enrolled 241 incl. 9 training cases (1 withdrew consent, 6 other); 2 Level ACDF enrolled 115 with no training cases (4 withdrew consent, 6 other)
Groups:
- 1 Level TDR: Cervical artificial disc (investigational device) at 1 level
- 1 Level ACDF: 1 level control procedure (ACDF)
- 2 Level TDR: Cervical artificial disc (investigational device) at 2 levels
- 2 Level ACDF: 2 level control procedure (ACDF)
Period: Overall Study
Arm/Group | 1 Level TDR | 1 Level ACDF | 2 Level TDR | 2 Level ACDF
Started | 164 | 81 | 225 | 105
24 mo | 156 | 75 | 221 | 99
Completed | 156 | 75 | 221 | 99
Not Completed | 8 | 6 | 4 | 6
Not completed — Lost to Follow-up | 8 | 6 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Level TDR | 1 Level ACDF | 2 Level TDR | 2 Level ACDF | Total
Number analyzed (Participants) | 164 | 81 | 225 | 105 | 575
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 161 | 80 | 222 | 101 | 564
  >=65 years | 3 | 1 | 3 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 45 | 112 | 45 | 288
  Male | 78 | 36 | 113 | 60 | 287
Region of Enrollment [Number; unit: participants]
  United States | 164 | 81 | 225 | 105 | 575

OUTCOME MEASURES:

1. Primary Outcome: Composite Definition of Study Success
Description: An individual subject in either treatment group was considered a success if the following criteria were met at 24 months:
  * Improvement in Neck Disability Index of at least 15/50 points in subjects with baseline Neck Disability Index scores of >= 30/50 points, or a 50% improvement in subjects with a baseline Neck Disability Score score of <30/50 where the Neck Disability Index is a measure designed to enable the physician to understand how much a subject's neck pain has affected his ability to manage everyday activities.
  * No study failures due to secondary surgical interventions at the index level
  * Absence of major complications defined as radiographic failure, neurologic failure, or failure by adverse event as adjudicated by the CEC
Time Frame: 2 Years
Population: includes study failures, per protocol, that are carried forward for overall success
Measure: Number; unit: percentage of subjects analyzed
Groups:
- 1 Level ACDF: control procedure (ACDF) at one level
- 2 Level ACDF: Cervical artificial disc (investigational device) at 2 levels compared with control procedure (ACDF) at two levels
- 2 Level TDR: control procedure (ACDF) at two levels
Arm/Group | 1 Level ACDF | 1 Level TDR | 2 Level ACDF | 2 Level TDR
Number analyzed (Participants) | 75 | 156 | 99 | 221
percentage of subjects analyzed | 65.3 | 73.7 | 37.4 | 69.7
Statistical Analysis 1: Comparison: 1 Level ACDF vs 1 Level TDR; 1 Level: Ho: pm-pc <=-0.1 (inferiority) Alternative hypothesis: Ha: pm - pc > -0.1 Where pm = the proportion of success in the Mobi-C group and the Pc = the proportion of success in the ACDF group; Test type: Non-Inferiority or Equivalence — The 95% one-sided confidence bound for testing non-inferiority using two proportion test with 10% non-inferiority margin; p = 0.0021, Farrington Manning
Statistical Analysis 2: Comparison: 2 Level ACDF vs 2 Level TDR; 2 Level: Ho: pm-pc <=-0.1 (inferiority) Alternative hypothesis: Ha: pm - pc > -0.1 Where pm = the proportion of success in the Mobi-C group and the Pc = the proportion of success in the ACDF group. 2 Level: Ho: pm-pc <= 0 (not superior) Alternative hypothesis: Ha: pm-pc >0 Where pm = the proportion of success in the Mobi-C group and the Pc = the proportion of success in the ACDF group; Test type: Non-Inferiority or Equivalence — The 95% one-sided confidence bound for testing non-inferiority using two proportioned test with a 10% non-inferiority margin; p < 0.0001, Farrington-Manning

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events are reported on all patients treated, including 24 surgical training subjects. Randomized total = 575, safety population total =599
Groups:
- 1 Level TDR Arm: Cervical artificial disc (investigational device) at 1 level
- 2 Level TDR Arm: Cervical artificial disc (investigational device) at 2 levels
Arm/Group | 1 Level TDR Arm | 1 Level ACDF Arm | 2 Level TDR Arm | 2 Level ACDF Arm
Serious Adverse Events (participants affected / at risk) | 32/179 | 21/81 | 56/234 | 34/105
Other Adverse Events (participants affected / at risk) | 170/179 | 75/81 | 209/234 | 100/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Level TDR Arm (N=179) | 1 Level ACDF Arm (N=81) | 2 Level TDR Arm (N=234) | 2 Level ACDF Arm (N=105)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 1 (1) | 0 (0) — All reported of AEs of cancer (malignancy or malignant tumor/neoplasm)
Anatomy/Technical Difficulty (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — Anatomy/Technical Difficulty includes Cervical - Study Surgery, Cervical - Non Study Surgery and Non Cervical
Cardiovascular (Cardiac disorders) | 4 (4) | 1 (1) | 7 (9) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — includes all deaths not related to the device - respiratory, cardiac, etc
Dysphagia/Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (2) | 2 (2) — includes all reported AEs of Dysphagia and other terms consistent with "difficulty swallowing" and all reported AEs of Dysphonia and other terms consistent with "voice change and/or disruption".
Gastrointestinal (Gastrointestinal disorders) | 5 (8) | 1 (2) | 3 (3) | 2 (2)
Heterotopic Ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Heterotopic Ossification includes Cervical - Index Level, Cervical - Adjacent Level and Non Cervical
Infection (Infections and infestations) | 3 (5) | 4 (6) | 6 (9) | 3 (4) — Infection includes Superficial Wound - Cervical, Deep Wound - Cervical, Other Wound - Non Study Surgery, both Systemic and Local
Malpositioned implant (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — includes misplaced screw, subsidence, a sub optimal or undesired position, regardless of causality. This is not mutually exclusive to surgeon error or sub-optimal placement of the original implant configuration.
Neck and/or Arm Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (4) | 10 (15) | 6 (8) — Neck and/or Arm Pain includes pain (and related pain terms) specific to neck (cervical spine) and arm pain (and related pain terms) specific to arm (spinal disorders are recorded elsewhere).
Neurological (Nervous system disorders) | 5 (8) | 3 (4) | 5 (5) | 5 (5) — Neurological including Upper Extremity - Sensory, motor, reflex; Lower Extremity - Sensory, motor, reflex; Upper & Lower Extremity - Sensory, motor, reflex; neck, back, spinal cord disturbance; gait disturbance, non specific and other
Non-union (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 1 (3) | 11 (14) — Non-Union includes non-union, cervical fusion failure, pseudoarthrosis, and pending non-unions as reported ; limited to study surgery related events of non-union.
Other (General disorders) | 6 (8) | 1 (1) | 12 (14) | 9 (13) — includes Blood/Lymphatic, Congenital/Genetic, Ear/Labyrinth, Endocrine, Eye, Immune, Metabolism/Nutrition, Musculoskeletal /CT, Benign Neoplasm, Nervous, Psychiatric, Repro, Skin, Vascular , Poisoning, Pregnancy, Social & surgical/Medical procedures
Other pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (4) | 10 (15) | 3 (3) — Other Pain including Shoulder, Back, Torso, Lower Extremity, Headache, Other
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (8) | 4 (4) | 7 (8) — Spinal Disorder including Cervical - Study Surgery, Cervical - Non Study Surgery and Non Cervical
Trauma (Social circumstances) | 4 (5) | 5 (8) | 7 (10) | 2 — includes falls, motor vehicle accidents, assault, injury, etc. This category includes both cervical and non-cervical AEs of Trauma.
Urogenital (Renal and urinary disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Upper Extremity Nerve Entrapment (Nervous system disorders) | 3 (3) | 1 (2) | 4 (5) | 0 (0) — including all reported AEs of Carpel Tunnel Syndrome and Cubital Tunnel Syndrome, including AEs directly attributed to Carpel Tunnel Syndrome or Cubital Tunnel Syndrome, as well as Carpal Tunnel surgery.
Wound Issue - Non-infection (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3) — including Hematoma, Hematoma Evacuation and CSF Leakage
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Level TDR Arm (N=179) | 1 Level ACDF Arm (N=81) | 2 Level TDR Arm (N=234) | 2 Level ACDF Arm (N=105)
Anatomy/Techical Difficulty (Surgical and medical procedures) | 11 (12) | 2 (4) | 9 (9) | 5 (5)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 1 (2) | 3 (3) | 1 (1)
Cardiovascular (Cardiac disorders) | 20 (26) | 10 (10) | 21 (29) | 10 (12)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia/Dysphonia (Respiratory, thoracic and mediastinal disorders) | 20 (26) | 17 (20) | 39 (43) | 24 (27)
Gastrointestinal (Gastrointestinal disorders) | 39 (60) | 15 (37) | 47 (97) | 32 (52)
Heterotopic Ossification (Musculoskeletal and connective tissue disorders) | 9 (10) | 4 (4) | 6 (6) | 1 (1)
Infection (Infections and infestations) | 33 (51) | 20 (28) | 56 (98) | 30 (50)
Malpositioned Implant (Surgical and medical procedures) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Neck and/or Arm Pain (Musculoskeletal and connective tissue disorders) | 101 (212) | 47 (98) | 102 (167) | 63 (111)
Neurological (Nervous system disorders) | 121 (401) | 52 (215) | 124 (426) | 78 (278)
Non-Union (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 1 (3) | 13 (18)
Other (General disorders) | 77 (114) | 33 (66) | 99 (189) | 58 (104)
Other Pain (Musculoskeletal and connective tissue disorders) | 102 (226) | 47 (144) | 131 (267) | 64 (132)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (8) | 19 (29) | 11 (12)
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 6 (7) | 10 (12) | 13 (18) | 13 (20)
Trauma (Social circumstances) | 47 (70) | 20 (38) | 52 (89) | 20 (36)
Upper Extremity Nerve Entrapment (Nervous system disorders) | 8 (9) | 4 (5) | 13 (16) | 6 (7)
Urogenital (Renal and urinary disorders) | 9 (11) | 9 (12) | 15 (23) | 10 (14)
Vascular Intraoperative (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound Issue -- Non-Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical site must submit to the Company, for review, any manuscripts, papers, summaries, abstracts, outlines or other media for publication at least 60 days before disclosure for the Company to review. The company has 30 days to review the proposed publication for any patentable subject matter or designated confidential information or confidential health information and by written notice to the site/PI identify such text so that the Company has time to file a patent application.